CLINICAL TRIAL: NCT00578110
Title: SBIR II Instrument for Glaucoma Early Detection and Monitoring
Brief Title: Instrument for Glaucoma Early Detection and Monitoring
Acronym: IGDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Synabridge Corporation (Industry)
Collaborators: Yale University (Other); University of Alabama at Birmingham (Other); University of Tennessee (Other)
Responsible Party: George Hu, President, Synabridge Corp.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPTH_DEV_GLAU_02; 1R43EY015015-01 (NIH); 1R43EY015015-02 (NIH); 1R43EY015015-03 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-20 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Glaucoma
Keywords: glaucoma VEP detection device diagnosis vision
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Glaucoma Patients
  Interventions: Device: Glaucoma Diagnosis, Name: Neucodia
- Group 2 (Experimental): Glaucoma suspects
  Interventions: Device: Glaucoma Diagnosis, Name: Neucodia
- Group 3 (Active Comparator): Controls
  Interventions: Device: Glaucoma Diagnosis, Name: Neucodia

INTERVENTIONS:
Device: Glaucoma Diagnosis, Name: Neucodia — Sensitivity and Specificity
  Other Names: NEUCODIA

SUMMARY:
To introduce a rapid and objective electrophysiological technique that can assess visual function in the magnocellular pathway, which is thought to be affected in early-stage glaucoma.

DETAILED DESCRIPTION:
The clinical study will evaluate a novel instrument designed to record visual evoked potentials elicited by stimuli determined in prior research (Greenstein et al., 1998; Badr et al., 2003) to drive select visual pathways that exhibit glaucomatous damage in an efficient and automated manner. The results obtained with this novel device will be compared with results obtained using an existing commercial device. Statistical results, sensitivity and specificity, will be generated for the assessment of the accuracy of the test to discriminate glaucoma patients from controls. Repeatability of the test will also be analyzed based on the test-retest results.

Visual evoked potential (VEP) is a measure of neural function in the eye and brain. Three skin electrodes are placed on the surface of the scalp to record the electrical activity from the brain while the subject is observing a flickering stimulus with isolated-check/dot pattern. The whole procedure is non-invasive and the risks are negligible.

Isolated-Check/dot Stimuli of about 10 Hz with luminance contrast of 10%, 15%, -10%, and -15% will be used to test each eye. Eight samples for each stimulus will be recorded. Each experimental run takes 2 seconds. The T-circ statistical method is performed to process the data, and the VEP signal to noise ratio (SNR) is calculated in order to obtain an optimized condition (stimulus and threshold) to separate glaucoma patients and normal group.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 - 75 years old
* Visual acuity: 20/30 or better

Exclusion Criteria:

* Eye disease other than glaucoma

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity | one year

SECONDARY OUTCOMES:
repeatability | one year

CONTACTS AND LOCATIONS:
Overall Officials: George Hu, Ph.D., Principal Investigator — Synabridge Corp.; James Tsai, M.D., Principal Investigator — Yale University; Max Forbes, M.D., Study Director — Columbia University; Vivienne Greenstein, Ph.D., Study Director — Columbia University; Eugenue Hartmann, Ph.D., Principal Investigator — University of Alabama at Birmingham; Peter Netland, M.D. Ph.D., Principal Investigator — University of Tennessee; Leo Pau Semes, O.D., Study Director — University of Alabama at Birmingham; Vance M Zemon, Ph.D., Study Director — Yeshiva University; Sarwat Salim, MD, Principal Investigator — University of Tennessee; Mark Swanson, OD, Study Director — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - School of Optometry, University of Alabama at Birmingham, Birmingham, Alabama
  - Yale Eye Center, Yale University, New Haven, Connecticut
  - Synabridge Corp., Raritan, New Jersey
  - Edward S. Harkness Eye Institute, Columbia University, New York, New York
  - Hamilton Eye Institute, The University of Tennessee, Memphis, Tennessee